CLINICAL TRIAL: NCT02756806
Title: A Clinical Evaluation of a Novel Multi-Wavelength Laser for Tattoo Removal
Brief Title: A Clinical Evaluation for Tattoo Removal
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change protocol to include multiple sites.
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-16-EN11
Record Dates: First submitted 2016-04-28; First posted 2016-04-29 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Tattoo Removal
Keywords: Tattoo removal, Picosecond Laser, Q-switched Laser

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Picosecond Q-switched Laser (Experimental): Treatment with investigational wavelengths of the Cutera enlighten laser for tattoo removal.
  Interventions: Device: Picosecond Q-switched laser

INTERVENTIONS:
Device: Picosecond Q-switched laser — Each subject will receive laser treatments with Enlighten laser
  Other Names: Enlighten

SUMMARY:
Evaluate safety and efficacy with the enlighten laser for tattoo removal.

DETAILED DESCRIPTION:
The purpose of this investigation is to evaluate the safety and efficacy of an investigational version of the Cutera enlighten laser for tattoo removal.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male, 18 to 65 years of age (inclusive).
* Fitzpatrick Skin Type I - VI (Appendix 3).
* Target tattoo contains single or multi-color ink, which includes blue and/or green.
* Target tattoos must be older than 1 year.
* Target tattoo not to exceed 12 square inches.
* Subject must be able to read, understand and sign the Informed Consent Form.
* Must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions.
* Wiling to cover tattoos with a bandage or clothing; and/or have very limited sun exposure and use an approved sunscreen of SPF 50 or higher on the treated area starting 2 to 4 weeks before the treatment and/or every day for the duration of the study, including the follow-up period.
* Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation, educational or marketing purposes.
* Agree to not undergo any other procedure(s) for tattoo removal during the study (as applicable).
* Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study, and no plans to become pregnant for the duration of the study.

Exclusion Criteria:

* Participation in a clinical trial of a drug or another device in the target area within 6 months prior to enrollment or during the study.
* Target tattoo contains only black ink.
* Target tattoo is a double tattoo where a first tattoo was covered with a second tattoo.
* History of allergic reaction to pigments following tattooing.
* History of allergy to local anesthetics.
* History of allergy to topical antibiotics.
* History of malignant tumors in the target area.
* Skin abnormalities in the target area, e.g., cuts, scrapes, wounds, scars, large moles.
* Pregnant and/or breastfeeding.
* Having an infection, dermatitis or a rash in the treatment area.
* Significant concurrent illness, such as diabetes mellitus or cardiovascular disease, e.g., uncontrolled hypertension.
* Suffering from coagulation disorders or taking prescription anticoagulation medications.
* History of keloid scarring, hypertrophic scarring or of abnormal wound healing.
* History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
* History of vitiligo, eczema, or psoriasis.
* History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.
* History of seizure disorders due to light.
* Any use of medication that is known to increase sensitivity to light according to Investigator's discretion.
* History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen
* History of radiation to the treatment area or undergoing systemic chemotherapy for the treatment of cancer.
* History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
* Systemic use of corticosteroid or isotretinoin within 6 months of study participation.
* Anytime in life, having used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus.
* Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
* Current smoker or history of smoking within 6 months of study participation.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-04; Primary Completion 2016-09-28 (Actual); Study Completion 2016-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Moldre, NP, Principal Investigator — Cutera Inc.
Locations (1):
- Cutera Research Center, Brisbane, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Picosecond Q-switched Laser
Started | 7
Completed | 2
Not Completed | 5
Not completed — Study terminated early | 5

BASELINE CHARACTERISTICS:
Groups:
- Picosecond Q-switched Laser: Treatment with investigational wavelengths of the Cutera enlighten laser for tattoo removal.
  Picosecond Q-switched laser: Each subject will receive up to 6 laser treatments.
Arm/Group | Picosecond Q-switched Laser
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: YEARS] | 45 [43 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Degree of Tattoo Clearing
Description: Degree of tattoo clearing at 12 weeks post-final treatment as assessed by independent blinded reviewers (Physician's Global Assessment of Improvement).
  Min=0; Max=4 Higher score indicate better tattoo clearing 4= Very Significant Clearing (>75%) 3 = Significant Clearing (51-75%) 2 = Moderate Clearing (26-50%)
  1 = Mild Clearing (5-25%) 0 = No Change (<5%)
Time Frame: 12-weeks post-final treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Picosecond Q-switched Laser
Number analyzed (Participants) | 2
score on a scale | 3 (0)

ADVERSE EVENTS:
Arm/Group | Picosecond Q-switched Laser
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Picosecond Q-switched Laser (N=7)
Frosting (Skin and subcutaneous tissue disorders) | 7
Erythema (Skin and subcutaneous tissue disorders) | 7
Edema (Skin and subcutaneous tissue disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No